CLINICAL TRIAL: NCT01908816
Title: An Open-label Extended Clinical Protocol of Ranibizumab to Evaluate Safety and Efficacy in Rare VEGF Driven Ocular Diseases.
Acronym: ECLIPSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002GFR02
Record Dates: First submitted 2013-07-20; First posted 2013-07-26 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Choroidal Neovascularization; Macular Edema; Glaucoma, Neovascular; Diabetic Retinopathy
MeSH Terms: conditions — Choroidal Neovascularization; Macular Edema; Glaucoma, Neovascular; Diabetic Retinopathy | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ranibizumab (Experimental): 0.5 mg ranibizumab applied in an individualized regimen as IVT injection of 0.05 mL.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — One injection of Ranibizumab 0.5 mg and retreatment according to disease activity and/or visual impairment on an as needed regimen (PRN)

SUMMARY:
The pupose of this study is to evaluate the safety and the efficacy of ranibizumab in rare VEGF driven ocular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Active choroidal neovascularization (CNV)
* Active macular edema (ME)
* Rubeosis iridis/neovascular glaucoma.
* Proliferative diabetic retinopathy requiring vitrectomy.

Exclusion Criteria:

* wet Age-related macular degeneration
* pathologic myopia
* pseudoxanthoma elasticum
* diabetic macular edema
* retinal vein occlusion
* < 18 years of age
* History of hypersensitivity to ranibizumab
* Use of any systemic anti-angiogenic drugs 3 months before inclusion
* Women of child-bearing potential and Pregnant or nursing (lactating) women.
* Active or suspected ocular infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2016-01-08 (Actual); Study Completion 2016-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- France (28):
  - Novartis Investigative Site, Bobigny, Seine Saint Denis
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Écully
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Mantes-la-Jolie
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Melun
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Jean
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Saitnt Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Vannes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: open-label, single arm study evaluating the safety of 0.5 mg ranibizumab. Patients received individualized ranibizumab intravitreal injections based on evidence of disease activity. The study was early terminated due to low recruitment that hampered to address the primary endpoint of the study
Groups:
- CNV (Choroidal Neovascularization); ME (Macular Edema); RI/NVG (Rubeosis Iridis and Neovacular Glaucoma): All patients received 0.5 mg ranibizumab IVT injection
- PDR/V: (Proliferative Diabetic Retinopathy requiring Vitrectomy). All patients received 0.5 mg ranibizumab IVT injection
Period: Overall Study
Arm/Group | CNV (Choroidal Neovascularization) | ME (Macular Edema) | RI/NVG (Rubeosis Iridis and Neovacular Glaucoma) | PDR/V
Started | 93 | 84 | 58 | 35
Completed | 0 | 0 | 0 | 0
Not Completed | 93 | 84 | 58 | 35
Not completed — Subject's no longer requires study drug | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 1 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 2
Not completed — Lost to Follow-up | 3 | 5 | 4 | 2
Not completed — Death | 1 | 0 | 7 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 13 | 1 | 0
Not completed — Early termination | 87 | 60 | 43 | 28

BASELINE CHARACTERISTICS:
Population: A total of 267 patients who received ranibizumab and had at least one post-baseline efficacy assessment were included in the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | CNV (Choroidal Neovascularization) | ME (Macular Edema) | RI/NVG (Rubeosis Iridis and Neovacular Glaucoma) | PDR/V | Total
Number analyzed (Participants) | 93 | 84 | 56 | 34 | 267
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (16.85) | 64.5 (13.99) | 70.9 (13.02) | 56.5 (9.86) | 59.7 (16.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 35 | 26 | 17 | 126
  Male | 45 | 49 | 30 | 17 | 141

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) for ocular and non-ocular events. Due to early termination, only descriptive analysis was conducted.
Time Frame: 24 months
Population: Safety population: all patients who received at least one application of study treatment and had at least one post-baseline safety assessment. The statement that a patient had no adverse events also constituted a safety assessment. All safety evaluations were carried out on the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CNV (Choroidal Neovascularization) | ME (Macular Edema) | RI/NVG (Rubeosis Iridis and Neovacular Glaucoma) | PDR/V
Number analyzed (Participants) | 93 | 84 | 58 | 35
Participants
  Non- serious adverse events | 2 | 21 | 1 | 0
  Serious adverse events | 11 | 15 | 31 | 14
  Death | 1 | 0 | 7 | 1

2. Secondary Outcome: Change From Baseline Best Corrected Visual Acuity (BCVA) for Patients With Choroidal Neovascularization (CNV) and Macular Edema (ME)
Description: BCVA change for diseases affecting the macular area either through CNV or ME. BCVA is tested using the ETDRS (Early Treatment Diabetic Retinopathy Study), the Snellen or Monoyer scales. The three scales are designed to measure visual acuity. ETDRS score is expressed in letter, Snellen and Monoyer score in fraction. BCVA assessment is presented in ETDRS after conversion if collected in Snellen or Monoyer. (Monoyer converted to Snellen = 2 x (Monoyer fraction) and Snellen converted to approximate ETDRS letters = 1x log(Snellen fraction). ETDRS letter score was transformed in logMAR unit for statistical analysis (- LogMAR = -(ETDRS-85)/50). The worse ETDRS letter score is 0 (logMAR 2.3) and the best ETDRS letter score is 100 (logMAR -0.3).
Time Frame: 3 months, 12 months
Population: Intent-to-treat population (ITT): all patients who received at least one application of study treatment and had at least one post-baseline efficacy assessment. The ITT population was the main analysis set for efficacy evaluations
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | CNV (Choroidal Neovascularization) | ME (Macular Edema)
Number analyzed (Participants) | 93 | 84
Letters
  3 Month: number analyzed (Participants) | 74 | 69
  3 Month | 7.3 (14.47) | 4.5 (11.61)
  12 Month: number analyzed (Participants) | 47 | 39
  12 Month | 5.7 (12.08) | 5.2 (16.46)

3. Secondary Outcome: Average Change of Neovascularization Extension for Patients With Neovascular Glaucoma
Description: The extent of iris neovascularization was assessed by iris photography and graded using the "Teich and Walsh grading system". This grading system measures the number of quadrant at iris pupillary zone or iris ciliary zone where iris neovascularization (NV) is observed.
  Grade 0 = "No iris vascularization", Grade 1= Less than 2 quadrants of NV at iris pupillary zone, Grade 2 = More than 2 quadrants of NV at iris pupillary zone, Grade 3 =Grade 2 + less than 3 quadrants of NV at iris ciliary zone and/or ectropion uveae; Grade 4 =More than 3 quadrants of NV at iris ciliary zone and/or ectropion uveae)
Time Frame: 3 month, 12 month
Population: as for outcome 2
Measure: Number; unit: Teich and Walsh grading
Groups:
- Ranibizumab 0.5 mg: All patients received 0.5 mg ranibizumab IVT injection
Arm/Group | Ranibizumab 0.5 mg
Number analyzed (Participants) | 56
Teich and Walsh grading
  3 Month,Grade 0: number analyzed (Participants) | 31
  3 Month,Grade 0 | 12
  3 Month, Grade 1: number analyzed (Participants) | 31
  3 Month, Grade 1 | 6
  3 Month, Grade 2: number analyzed (Participants) | 31
  3 Month, Grade 2 | 8
  3 Month, Grade 3: number analyzed (Participants) | 31
  3 Month, Grade 3 | 3
  3 Month, Grade 4: number analyzed (Participants) | 31
  3 Month, Grade 4 | 2
  12 Month, Grade 0: number analyzed (Participants) | 25
  12 Month, Grade 0 | 11
  12 Month, Grade 1: number analyzed (Participants) | 25
  12 Month, Grade 1 | 4
  12 Month, Grade 2: number analyzed (Participants) | 25
  12 Month, Grade 2 | 2
  12 Month, Grade 3: number analyzed (Participants) | 25
  12 Month, Grade 3 | 4
  12 Month, Grade 4: number analyzed (Participants) | 25
  12 Month, Grade 4 | 4

4. Secondary Outcome: Proportion of Patient With Vitreous Cavity Hemorrhage Occurrence for Patient With Proliferative Retinopathy
Description: Occurrence of postoperative vitreous cavity hemorrhage
Time Frame: 3 months, 12 month
Population: Intent-to-treat population (ITT): all patients who received at least one application of study treatment and had at least one post-baseline efficacy assessment. The ITT population was the main analysis set for efficacy evaluations. (n) is the number of participants with an observed value
Measure: Number; unit: Participants
Arm/Group | PDR/V
Number analyzed (Participants) | 34
Participants
  3 Month Absent: number analyzed (Participants) | 17
  3 Month Absent | 14
  3 Month Present: number analyzed (Participants) | 17
  3 Month Present | 3
  12 Month Absent: number analyzed (Participants) | 13
  12 Month Absent | 12
  12 Month Present: number analyzed (Participants) | 13
  12 Month Present | 1

5. Secondary Outcome: Mean Change From Baseline in Change in Central Retinal Thickness for Patients With CNV (Choroidal Neovascularization) and ME (Macular Edema)"
Description: CRT in micrometers assessed by Optical Tomography (OCT) at each single study visit. A reduction is thickness indicates an improvement is the lesion area
Time Frame: 3 months, 12 month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | CNV (Choroidal Neovascularization) | ME (Macular Edema)
Number analyzed (Participants) | 93 | 84
μm
  3 Month: number analyzed (Participants) | 74 | 67
  3 Month | -54.4 (104.55) | -84.4 (178.28)
  12 Month: number analyzed (Participants) | 45 | 40
  12 Month | -56.4 (69.82) | -102.0 (220)

6. Secondary Outcome: Proportion of Patients With Angiographic Leakage
Description: Angiography was taken via fluorescein angiography. Any increases of angiographic leakage was counted between baseline and month 3. Also any decreases of angiographic leakage was counted between baseline and 3 month.
Time Frame: 3 months, 12 month
Population: Intent-to-treat population (ITT): all patients who received at least one application of study treatment and had at least one post-baseline efficacy assessment. The ITT population was the main analysis set for efficacy evaluations. The (n) represent the number of assessed value.
Measure: Number; unit: Participants
Arm/Group | CNV (Choroidal Neovascularization) | ME (Macular Edema) | PDR/V
Number analyzed (Participants) | 93 | 84 | 34
Participants
  3 Month Absent: number analyzed (Participants) | 6 | 6 | 1
  3 Month Absent | 3 | 3 | 1
  3 Month Present: number analyzed (Participants) | 6 | 6 | 1
  3 Month Present | 3 | 3 | 0
  12 Month Absent: number analyzed (Participants) | 5 | 1 | 0
  12 Month Absent | 3 | 1 |
  12 Month Present: number analyzed (Participants) | 5 | 1 | 0
  12 Month Present | 2 | 0 |

7. Secondary Outcome: Ranibizumab Injection
Description: Number of ranibizumab injections needed by decreased visual acuity and/or increasing retinal thickness in 3 months of observation period
Time Frame: 3 months, 12 month
Population: Safety set population: all patients who received at least one application of study treatment and had at least one post-baseline safety assessment. The statement that a patient had no adverse events also constituted a safety assessment. All safety evaluations were carried out on the safety population.
Measure: Mean (Standard Deviation); unit: Number of injections
Arm/Group | CNV (Choroidal Neovascularization) | ME (Macular Edema) | RI/NVG (Rubeosis Iridis and Neovacular Glaucoma) | PDR/V
Number analyzed (Participants) | 93 | 84 | 58 | 35
Number of injections
  3 Month: number analyzed (Participants) | 75 | 70 | 34 | 17
  3 Month | 2.5 (1.03) | 2.7 (0.88) | 1.7 (0.79) | 1.6 (1.0)
  12 Month: number analyzed (Participants) | 44 | 38 | 21 | 14
  12 Month | 3.8 (2.34) | 3.9 (2.17) | 3.0 (1.96) | 1.7 (1.44)

ADVERSE EVENTS:
Time Frame: up to 3 years
Description: AE additional description
Groups:
- Choroidal Neovascularization: Choroidal neovascularization
- Macular Edema: Macular edema
- Rubeosis Iridis/ Neovascular Glaucoma: Rubeosis iridis/ Neovascular glaucoma
- Proliferative Diabetic Retinopathy Requiring Vitrectomy: Proliferative diabetic retinopathy requiring vitrectomy
Arm/Group | Choroidal Neovascularization | Macular Edema | Rubeosis Iridis/ Neovascular Glaucoma | Proliferative Diabetic Retinopathy Requiring Vitrectomy
All-Cause Mortality (participants affected / at risk) | 1/93 | 0/84 | 7/58 | 1/35
Serious Adverse Events (participants affected / at risk) | 11/93 | 15/84 | 31/58 | 14/35
Other Adverse Events (participants affected / at risk) | 46/93 | 66/84 | 40/58 | 21/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Choroidal Neovascularization (N=93) | Macular Edema (N=84) | Rubeosis Iridis/ Neovascular Glaucoma (N=58) | Proliferative Diabetic Retinopathy Requiring Vitrectomy (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 4 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Anterior chamber fibrin (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Blindness (Both eyes) (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Contralateral eye) (Eye disorders) | 0 | 2 | 1 | 0
Cataract (Study eye) (Eye disorders) | 0 | 1 | 0 | 1
Glaucoma (Contralateral eye) (Eye disorders) | 0 | 0 | 0 | 1
Glaucoma (Study eye) (Eye disorders) | 0 | 0 | 2 | 1
Macular detachment (Both eyes) (Eye disorders) | 0 | 0 | 0 | 1
Macular fibrosis (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Ocular hypertension (Both eyes) (Eye disorders) | 0 | 0 | 1 | 0
Ocular hypertension (Study eye) (Eye disorders) | 1 | 1 | 7 | 0
Retinal artery occlusion (Both eyes) (Eye disorders) | 0 | 0 | 0 | 1
Retinal detachment (Study eye) (Eye disorders) | 0 | 0 | 3 | 1
Retinal pigment epithelial tear (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Retinal tear (Study eye) (Eye disorders) | 0 | 0 | 0 | 1
Visual acuity reduced (Both eyes) (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 0 | 1 | 1
Vitreous adhesions (Contralateral eye) (Eye disorders) | 0 | 0 | 0 | 1
Vitreous adhesions (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Vitreous haemorrhage (Contralateral eye) (Eye disorders) | 0 | 0 | 2 | 0
Vitreous haemorrhage (Study eye) (Eye disorders) | 0 | 2 | 2 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal dysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Drug ineffective (Study eye) (General disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Corneal abscess (Study eye) (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Syphilis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intraocular pressure increased (Study eye) (Investigations) | 0 | 1 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Choroid melanoma (Study eye) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Akinesia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephroangiosclerosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Arterial disorder (Vascular disorders) | 0 | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Choroidal Neovascularization (N=93) | Macular Edema (N=84) | Rubeosis Iridis/ Neovascular Glaucoma (N=58) | Proliferative Diabetic Retinopathy Requiring Vitrectomy (N=35)
Cataract (Study eye) (Eye disorders) | 0 | 3 | 1 | 0
Conjunctival haemorrhage (Study eye) (Eye disorders) | 0 | 4 | 0 | 1
Dry eye (Study eye) (Eye disorders) | 0 | 2 | 2 | 0
Eye pain (Study eye) (Eye disorders) | 6 | 5 | 7 | 3
Eye pruritus (Study eye) (Eye disorders) | 2 | 1 | 1 | 0
Ocular hyperaemia (Study eye) (Eye disorders) | 1 | 0 | 1 | 1
Ocular hypertension (Study eye) (Eye disorders) | 0 | 0 | 2 | 3
Punctate keratitis (Study eye) (Eye disorders) | 1 | 0 | 1 | 1
Ulcerative keratitis (Study eye) (Eye disorders) | 0 | 1 | 2 | 2
Vision blurred (Study eye) (Eye disorders) | 2 | 1 | 0 | 2
Visual acuity reduced (Contralateral eye) (Eye disorders) | 2 | 0 | 0 | 1
Visual acuity reduced (Study eye) (Eye disorders) | 3 | 3 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 3 | 0
Drug ineffective (Study eye) (General disorders) | 3 | 27 | 1 | 0
Fatigue (General disorders) | 2 | 3 | 4 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 0 | 1
Conjunctivitis (Both eyes) (Infections and infestations) | 1 | 1 | 0 | 1
Conjunctivitis (Study eye) (Infections and infestations) | 1 | 0 | 1 | 1
Influenza (Infections and infestations) | 4 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Inappropriate schedule of drug administration (Study eye) (Injury, poisoning and procedural complications) | 11 | 21 | 4 | 1
Incorrect product storage (Study eye) (Injury, poisoning and procedural complications) | 4 | 6 | 1 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 4 | 0 | 0
Headache (Nervous system disorders) | 7 | 4 | 2 | 0
Depression (Psychiatric disorders) | 0 | 1 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 2 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0
Allergic keratitis (Study eye) (Eye disorders) | 0 | 0 | 0 | 1
Anterior chamber fibrin (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Blepharitis (Both eyes) (Eye disorders) | 1 | 0 | 1 | 0
Blepharitis (Contralateral eye) (Eye disorders) | 1 | 0 | 1 | 0
Blepharospasm (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Both eyes) (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Contralateral eye) (Eye disorders) | 0 | 0 | 1 | 0
Cataract subcapsular (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Chalazion (Contralateral eye) (Eye disorders) | 0 | 0 | 1 | 0
Choroidal neovascularisation (Contralateral eye) (Eye disorders) | 1 | 0 | 0 | 0
Choroiditis (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Contralateral eye) (Eye disorders) | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Both eyes) (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Study eye) (Eye disorders) | 1 | 1 | 0 | 0
Conjunctival ulcer (Study eye) (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis allergic (Both eyes) (Eye disorders) | 1 | 1 | 0 | 0
Corneal perforation (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Cystoid macular oedema (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Both eyes) (Eye disorders) | 1 | 1 | 0 | 0
Eczema eyelids (Contralateral eye) (Eye disorders) | 0 | 1 | 0 | 0
Exophthalmos (Both eyes) (Eye disorders) | 0 | 1 | 0 | 0
Eye allergy (Both eyes) (Eye disorders) | 0 | 1 | 0 | 0
Eye discharge (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Eye haemorrhage (Study eye) (Eye disorders) | 0 | 0 | 2 | 0
Eye inflammation (Study eye) (Eye disorders) | 1 | 0 | 0 | 1
Eye irritation (Both eyes) (Eye disorders) | 2 | 0 | 0 | 0
Eye irritation (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Eye oedema (Study eye) (Eye disorders) | 0 | 0 | 0 | 1
Eye pain (Both eyes) (Eye disorders) | 0 | 0 | 1 | 1
Eye pain (Contralateral eye) (Eye disorders) | 0 | 0 | 1 | 0
Eye pruritus (Both eyes) (Eye disorders) | 1 | 0 | 0 | 1
Eye ulcer (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Eyelid cyst (Contralateral eye) (Eye disorders) | 1 | 0 | 0 | 0
Eyelid irritation (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Eyelid myoclonus (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Eyelid pain (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Eyelid ptosis (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Foreign body sensation in eyes (Both eyes) (Eye disorders) | 0 | 1 | 0 | 0
Foreign body sensation in eyes (Contralateral eye) (Eye disorders) | 1 | 0 | 0 | 0
Foreign body sensation in eyes (Study eye) (Eye disorders) | 0 | 0 | 1 | 1
Glare (Study eye) (Eye disorders) | 1 | 1 | 0 | 0
Glaucoma (Both eyes) (Eye disorders) | 0 | 0 | 1 | 0
Iridocyclitis (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Iris neovascularisation (Contralateral eye) (Eye disorders) | 0 | 0 | 1 | 0
Keratitis (Study eye) (Eye disorders) | 0 | 1 | 0 | 1
Lacrimation increased (Both eyes) (Eye disorders) | 0 | 0 | 0 | 1
Macular fibrosis (Study eye) (Eye disorders) | 2 | 0 | 0 | 0
Macular oedema (Study eye) (Eye disorders) | 1 | 1 | 0 | 0
Metamorphopsia (Study eye) (Eye disorders) | 2 | 0 | 0 | 0
Ocular discomfort (Contralateral eye) (Eye disorders) | 0 | 0 | 0 | 1
Ocular discomfort (Study eye) (Eye disorders) | 0 | 0 | 2 | 0
Ocular hypertension (Both eyes) (Eye disorders) | 0 | 1 | 1 | 0
Ocular hypertension (Contralateral eye) (Eye disorders) | 1 | 0 | 0 | 0
Photophobia (Both eyes) (Eye disorders) | 1 | 0 | 0 | 0
Photophobia (Contralateral eye) (Eye disorders) | 0 | 0 | 0 | 1
Photophobia (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Photopsia (Both eyes) (Eye disorders) | 1 | 0 | 0 | 0
Photopsia (Contralateral eye) (Eye disorders) | 1 | 0 | 0 | 0
Photopsia (Study eye) (Eye disorders) | 1 | 0 | 0 | 1
Punctate keratitis (Contralateral eye) (Eye disorders) | 0 | 0 | 1 | 0
Retinal detachment (Study eye) (Eye disorders) | 1 | 1 | 0 | 0
Retinal haemorrhage (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Retinal neovascularisation (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Retinal oedema (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Retinal pigment epithelial tear (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Retinal pigment epitheliopathy (Both eyes) (Eye disorders) | 1 | 0 | 0 | 0
Uveitis (Both eyes) (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Both eyes) (Eye disorders) | 0 | 0 | 2 | 0
Visual acuity reduced (Both eyes) (Eye disorders) | 0 | 1 | 0 | 1
Visual impairment (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Both eyes) (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Contralateral eye) (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Study eye) (Eye disorders) | 1 | 1 | 0 | 0
Vitreous haemorrhage (Study eye) (Eye disorders) | 0 | 0 | 0 | 1
Vitritis (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 1 | 0
Injection site ulcer (Study eye) (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Secretion discharge (Study eye) (General disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Eye infection (Study eye) (Infections and infestations) | 0 | 1 | 0 | 0
Genital infection female (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Infected bite (Infections and infestations) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural infection (Study eye) (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Conjunctival laceration (Study eye) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyphaema (Study eye) (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Incorrect product storage (Contralateral eye) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Intraocular pressure increased (Contralateral eye) (Investigations) | 0 | 1 | 0 | 0
Intraocular pressure increased (Study eye) (Investigations) | 0 | 1 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 2 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lymphoma cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Visual field defect (Study eye) (Nervous system disorders) | 1 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
As the study was early terminated, no conclusion could be drawn from this study. The data should be interpreted with cautious as less than half of the patients included in the study (47.0%) completed the visit at Month 12.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.